## Effects of intensified oral P2Y12 inhibition on elevated fibrin-platelet clot strength in patients with acute coronary syndromes (TEGCOR Study)

## **Principal Investigator:**

Rolf P. Kreutz, M.D. Krannert Institute of Cardiology 1701 N. Senate Blvd, ME-400 Indianapolis, IN 46202

## Statistical Analysis Plan

Comparison of clot strength measured by Thrombelastography in whole blood (TEG-MA) will be made with 2-sided Student's T-test after reloading of clopidogrel or prasugrel at 16-24 hours. Comparison of outcome events (death, recurrent myocardial infarction, recurrent unstable angina, repeat coronary intervention up to 6 months) will be made by Chi-Square test. All tests are performed two-sided with p<0.05 as significance threshold.